CLINICAL TRIAL: NCT06250660
Title: The Effectiveness of an Intervention Based on the Consumption of Fresh Strawberries From the Huelva Region on Menstrual Pain and Menstrual Distress in Young University Students
Brief Title: The Effectiveness of an Intervention of Fresh Strawberries on Menstrual Pain and Menstrual Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynthia del Rocío Márquez Beltrán (Other)
Collaborators: University of Huelva (Other)
Responsible Party: Sponsor-Investigator, Cynthia del Rocío Márquez Beltrán, PHD Student. Associate researcher. Nurse., University of Huelva
Organization: University of Huelva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PFH-1123
Record Dates: First submitted 2024-01-26; First posted 2024-02-09 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Primary Dysmenorrhea; Menstrual Pain; Menstrual Distress (Dysmenorrhea)
Keywords: strawberry; primary dysmenorrhea; menstrual distress; pelvic pain; menstruation disturbance
MeSH Terms: conditions — Dysmenorrhea; Pelvic Pain; Menstruation Disturbances

STUDY DESIGN:
Intervention Model Description: Women who meet the inclusion criteria will be divided into two groups. There will be an intervention group, corresponding to the intake of strawberry and a control group. Participants will be randomly assigned to each group, the randomization will be 1:1, so there will be the same number of participants in each of the two groups. The intervention group will receive the corresponding amount of strawberries and the control group will continue with their usual diet and treatment for dysmenorrhea.
Masking Description: The assignment to each group will be blind. It will be done through a computer application, which assigns random numbers to each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in the comparison group will not have intervention and will not receive strawberry supplements, they will follow their conventional treatment and their usual diet. They will be evaluated before the start of the intervention, one month and two months after the intervention.
- Strawberry intervention with Fortuna variety (Experimental): This group will receive an intake of strawberries of the Fortuna variety. The participants of this group will have to eat 250 g of this strawberry variety per day for 1 month.
  All participants in the intervention group will be invited to participate in focus groups once the intervention has ended, in order to learn about their experiences during it.
  They will be evaluated before the start of the intervention, one month and two months after the intervention.
  Interventions: Dietary Supplement: Strawberry Intervention

INTERVENTIONS:
Dietary Supplement: Strawberry Intervention — This is an intervention based on the intake of strawberry, specifically the "Fortuna" variety. This intervention is based on the intake of 250 g of fresh strawberries per day for a month. The amount and duration of strawberry intake has been consulted in other studies carried out with strawberries.
  Arms: Strawberry intervention with Fortuna variety

SUMMARY:
The purpose of this project is to know the effectiveness of an intervention based on the consumption of fresh strawberries from the Huelva region on menstrual pain and menstrual distress in young university students with primary dysmenorrhea, compared to a control group of students.

The participants with dysmenorrhea will be divided into two groups, the assignment will be random to the intervention group with strawberry intake for a month and comparing its effect with de control group. The results of the evaluations carried out prior, to the month and 2 months of the intervention will be compared.

DETAILED DESCRIPTION:
Dysmenorrhea is a prevalent problem among women of childbearing age; previous studies carried out among young university students have identified that it affects 74% of them. Dysmenorrhea can also be accompanied by the well-known menstrual distress, which has been estimated to affect between 75 and 94% of women. The symptoms included in menstrual distress are diverse, including irritability, nausea, vomiting, abdominal pain, general weakness or fatigue, among others. Dysmenorrhea and distress have a significant impact on the lives of women who suffer from it, affecting their social life, quality of life and academic and work performance.

The methods that women use to relieve dysmenorrhea are usually pharmacological, with NSAIDs (Non Steroidal Anti-Inflammatory Drugs) and hormonal contraceptives, but these are not free of adverse effects, so more and more studies are investigating non-pharmacological methods to relieve pain. Menstrual distress is also being included as an object of study.

A healthy lifestyle has been shown to be beneficial in relieving primary dysmenorrhoea. In particular, exercise and eating at least 2 pieces of fruit per day have been identified as protective habits.

Most of the studies that evaluate food intake in women with dysmenorrhea are observational and the few clinical trials that exist are with small samples. Strawberries are rich in flavonoids and phenolic acids, giving them anti-inflammatory and antioxidant properties. Studies carried out with strawberries have shown their benefits against chronic inflammatory and cardiovascular diseases. For these reasons, it is necessary a clinical trial to evaluate the benefits of strawberry in relieving dysmenorrhea and menstrual distress.

Carrying out a clinical trial with strawberries is a challenge. Firstly, there is no consensus on the optimal dose that should be ingested to influence health biomarkers. On the other hand, the use of fresh strawberries involves a significant cost, in addition to the fact that it is a seasonal fruit, which is why the most of trials with strawberries are carried out with freeze-dried strawberry powder.

The aim of this study is to analyze the benefits of strawberry consumption in relieving menstrual pain using the VAS (Visual Analogue Scale) scale and menstrual distress using the MEDI-Q scale, previously validated in Spanish in a previous phase of the study in female university students. The results obtained will be compared between the intervention group belonging to the intake of strawberry (specifically the "Fortuna" variety) and with a control group that will continue with their usual diet during the same period of time. They will be evaluated previously, one month and two months after receiving the intervention. The project has been approved by the Andalusian Ethics and Research Committee.

For the design of the clinical trial, previous studies on food intake and dysmenorrhea, as well as studies on the health benefits of strawberries, have been taken into account.

The "Fortuna" strawberry variety will be provided by the association Fres Huelva and must be eaten daily for a month. Participants will be provided with a menstrual diary in order to avoid forgetfulness bias. Participants who are part of the intervention group will be invited to participate in focus groups in order to know about their experiences during the trial.

Our hypothesis is that women who regularly consume strawberries in their diet will improve their pain intensity and levels of menstrual distress, as well as other symptoms associated with dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Suffer menstrual pain at least 1 time in the last 6 months or 3 times in the last year
* Without a history of diagnosed gynecological pathology
* Not taking hormonal contraception
* Being enrolled at the University of Huelva for the academic year 2023/2024

Exclusion Criteria:

* Those who do not meet the inclusion criteria
* Being in the process of mobility during the months of study
* Have had an abortion
* Suffer from a problem that requires limiting the consumption of fruit or strawberries in their diet
* Suffer from a chronic disease that causes pain

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change from baseline pain intensity at 1 month and 2 months.
  Pain intensity will be evaluated with the Visual Analog Scale (VAS). This is a self-administered, single-item measurement scale. Located on a horizontal or vertical line 10 cm (100mm) long, whose values range from 0 ("no pain") to 10 ("the worst pain imaginable"). Participants will be asked to write down the maximum perceived pain during the first 3 days of menstruation.
Distress menstrual | Change from baseline distress menstrual at 1 month and 2 months.
  Menstrual distress will be assessed using the MEDI-Q scale, which will be validated in Spanish in a previous phase of this study. This questionnaire evaluates symptoms in the premenstrual, menstrual and intermenstrual phases through a total of 25 items. The score ranges between 0 (absence of symptoms that cause distress during menstruation in the last year) and 125 (presence of all symptoms in more than half of menstruations in the last 12 months).

SECONDARY OUTCOMES:
Changes in Quality of life | Baseline, 1 month and 2 months.
  To assess quality of life, EuroQol-5D (EQ-5D) will be used. It is an element for measuring HRQoL (health-related quality of life) that measures 5 dimensions of health (mobility, personal care, usual activities, pain and discomfort and, finally, anxiety and depression). In the first part, the participant must evaluate their health status through the dimensions, the second part must evaluate their health status through a visual analog scale from 0 (worst imaginable health status) to 100 (best imaginable health status).
Anxiety State and Anxiety Trait | Baseline, 1 month and 2 months.
  Anxiety will be measured through the Spanish version of the State/Trait Anxiety Inventory (STAI), made up of the Anxiety/State and Anxiety/Trait scales, with 20 items each and a Likert-type response from 0 (not at all) to 3 (very much), obtaining a total score between 0 and 60. A higher score indicates a higher level of anxiety.
Perceived well-being | Baseline, 1 month and 2 months.
  Well-being will be measured with the Spanish version of the Warwick-Edinburgh Mental Well-being Scale (EBMWE). This scale consists of 14 items, with a Likert-type response option from 1 to 5. With a total score range between 14 and 70, a higher score indicates greater mental well-being.
Sleep quality | Baseline, 1 month and 2 months.
  Sleep quality will be measured with the Pittsburgh Sleep Quality Index (PSQI). It is a self-report scale to assess sleep quality divided into 7 parts with 19 items, associated in 10 questions, each of which is scored between 0 (ease) and 3 (severe difficulty). The total score ranges from 0 (ease of sleeping) to 21 (difficulty in all areas).
Changes amount of bleeding | Baseline, 1 month and 2 months.
  Changes in the amount of bleeding will be measured through questions about the number of sanitary towels at day in relation to the last menstruation.
Changes menstrual issues | Baseline, 1 month and 2 months.
  Menstrual issues will be assessed through questions about days of menstruation, and length of cycle (in days) in relation to the last menstruation.
Changes in menstrual pain management | Baseline, 1 month and 2 months.
  Questions will be asked to know the method used to relieve menstrual pain; in the case of pharmacological pain relief, the dose and type of drug, and the effectiveness of the method will be asked.
Changes in absenteeism and presenteeism days | Baseline, 1 month and 2 months.
  Absenteeism and presenteeism will be consulted, through questions regarding the number of days that absenteeism or presenteeism has occurred in relation to the last menstruation.
The impact on daily and academic activities | Baseline, 1 month and 2 months.
  The impact on daily and academic activities will be evaluated with specific questions that will be answered on a scale of 0-10 (where 0 is not having a limitation and 10 is the impossibility of doing it) in relation to different situations and activities with respect to the last menstruation

CONTACTS AND LOCATIONS:
Overall Officials: Elia Fernández Martínez, PHD, Study Director — Teacher and Researcher
Locations (1):
- Universidad de Huelva, Huelva, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armour M, Parry K, Manohar N, Holmes K, Ferfolja T, Curry C, MacMillan F, Smith CA. The Prevalence and Academic Impact of Dysmenorrhea in 21,573 Young Women: A Systematic Review and Meta-Analysis. J Womens Health (Larchmt). 2019 Aug;28(8):1161-1171. doi: 10.1089/jwh.2018.7615. Epub 2019 Jun 6. PMID 31170024
- [Background] Abreu-Sanchez A, Parra-Fernandez ML, Onieva-Zafra MD, Ramos-Pichardo JD, Fernandez-Martinez E. Type of Dysmenorrhea, Menstrual Characteristics and Symptoms in Nursing Students in Southern Spain. Healthcare (Basel). 2020 Aug 26;8(3):302. doi: 10.3390/healthcare8030302. PMID 32858887
- [Background] Cholbeigi E, Rezaienik S, Safari N, Lissack K, Griffiths MD, Alimoradi Z. Are health promoting lifestyles associated with pain intensity and menstrual distress among Iranian adolescent girls? BMC Pediatr. 2022 Oct 5;22(1):574. doi: 10.1186/s12887-022-03639-x. PMID 36199045
- [Background] Chen HM, Wang HH, Chiu MH, Hu HM. Effects of acupressure on menstrual distress and low back pain in dysmenorrheic young adult women: an experimental study. Pain Manag Nurs. 2015 Jun;16(3):188-97. doi: 10.1016/j.pmn.2014.06.002. Epub 2014 Aug 28. PMID 25175554
- [Background] Matthewman G, Lee A, Kaur JG, Daley AJ. Physical activity for primary dysmenorrhea: a systematic review and meta-analysis of randomized controlled trials. Am J Obstet Gynecol. 2018 Sep;219(3):255.e1-255.e20. doi: 10.1016/j.ajog.2018.04.001. Epub 2018 Apr 7. PMID 29630882
- [Background] Bajalan Z, Alimoradi Z, Moafi F. Nutrition as a Potential Factor of Primary Dysmenorrhea: A Systematic Review of Observational Studies. Gynecol Obstet Invest. 2019;84(3):209-224. doi: 10.1159/000495408. Epub 2019 Jan 10. PMID 30630172
- [Background] Cassioli E, Rossi E, Melani G, Faldi M, Rellini AH, Wyatt RB, Oester C, Vannuccini S, Petraglia F, Ricca V, Castellini G. The menstrual distress questionnaire (MEDI-Q): reliability and validity of the English version. Gynecol Endocrinol. 2023 Jun 19;39(1):2227275. doi: 10.1080/09513590.2023.2227275. PMID 37356456
- [Background] Vannuccini S, Rossi E, Cassioli E, Cirone D, Castellini G, Ricca V, Petraglia F. Menstrual Distress Questionnaire (MEDI-Q): a new tool to assess menstruation-related distress. Reprod Biomed Online. 2021 Dec;43(6):1107-1116. doi: 10.1016/j.rbmo.2021.08.029. Epub 2021 Oct 26. PMID 34753680
- [Background] Fernandez-Martinez E, Abreu-Sanchez A, Velarde-Garcia JF, Iglesias-Lopez MT, Perez-Corrales J, Palacios-Cena D. Living with Restrictions. The Perspective of Nursing Students with Primary Dysmenorrhea. Int J Environ Res Public Health. 2020 Nov 17;17(22):8527. doi: 10.3390/ijerph17228527. PMID 33212985
- [Background] Fernandez-Martinez E, Abreu-Sanchez A, Perez-Corrales J, Ruiz-Castillo J, Velarde-Garcia JF, Palacios-Cena D. Living with Pain and Looking for a Safe Environment: A Qualitative Study among Nursing Students with Dysmenorrhea. Int J Environ Res Public Health. 2020 Sep 13;17(18):6670. doi: 10.3390/ijerph17186670. PMID 32933209
- [Background] Rodrigues AC, Gala S, Neves A, Pinto C, Meirelles C, Frutuoso C, Vitor ME. [Dysmenorrhea in adolescents and young adults: prevalence, related factors and limitations in daily living]. Acta Med Port. 2011 Dec;24 Suppl 2:383-88; quiz 389-92. Epub 2011 Dec 31. Portuguese. PMID 22849926
- [Background] Vannuccini S, Clemenza S, Cassioli E, Rossi E, Castellini G, Ricca V, Petraglia F. Uterine Fibroids, Perceived Stress, and Menstrual Distress: a Key Role of Heavy Menstrual Bleeding. Reprod Sci. 2023 May;30(5):1608-1615. doi: 10.1007/s43032-022-01126-3. Epub 2022 Dec 5. PMID 36471219
- [Background] Parra-Fernandez ML, Onieva-Zafra MD, Abreu-Sanchez A, Ramos-Pichardo JD, Iglesias-Lopez MT, Fernandez-Martinez E. Management of Primary Dysmenorrhea among University Students in the South of Spain and Family Influence. Int J Environ Res Public Health. 2020 Aug 1;17(15):5570. doi: 10.3390/ijerph17155570. PMID 32752254
- [Background] Fernandez-Martinez E, Perez-Corrales J, Palacios-Cena D, Abreu-Sanchez A, Iglesias-Lopez MT, Carrasco-Garrido P, Velarde-Garcia JF. Pain management and coping strategies for primary dysmenorrhea: A qualitative study among female nursing students. Nurs Open. 2022 Jan;9(1):637-645. doi: 10.1002/nop2.1111. Epub 2021 Oct 30. PMID 34719126
- [Background] Giampieri F, Alvarez-Suarez JM, Battino M. Strawberry and human health: effects beyond antioxidant activity. J Agric Food Chem. 2014 May 7;62(18):3867-76. doi: 10.1021/jf405455n. Epub 2014 Feb 3. PMID 24450925
- [Background] Huang L, Xiao D, Zhang X, Sandhu AK, Chandra P, Kay C, Edirisinghe I, Burton-Freeman B. Strawberry Consumption, Cardiometabolic Risk Factors, and Vascular Function: A Randomized Controlled Trial in Adults with Moderate Hypercholesterolemia. J Nutr. 2021 Jun 1;151(6):1517-1526. doi: 10.1093/jn/nxab034. PMID 33758944
- [Background] O'Doherty AF, Jones HS, Sathyapalan T, Ingle L, Carroll S. The Effects of Acute Interval Exercise and Strawberry Intake on Postprandial Lipemia. Med Sci Sports Exerc. 2017 Nov;49(11):2315-2323. doi: 10.1249/MSS.0000000000001341. PMID 29045326
- [Background] Ezzat-Zadeh Z, Henning SM, Yang J, Woo SL, Lee RP, Huang J, Thames G, Gilbuena I, Tseng CH, Heber D, Li Z. California strawberry consumption increased the abundance of gut microorganisms related to lean body weight, health and longevity in healthy subjects. Nutr Res. 2021 Jan;85:60-70. doi: 10.1016/j.nutres.2020.12.006. Epub 2020 Dec 5. PMID 33450667
- [Background] Nikkhah S, Dolatian M, Naghii MR, Zaeri F, Taheri SM. Effects of boron supplementation on the severity and duration of pain in primary dysmenorrhea. Complement Ther Clin Pract. 2015 May;21(2):79-83. doi: 10.1016/j.ctcp.2015.03.005. Epub 2015 Apr 4. PMID 25906949
- [Background] Herdman M, Badia X, Berra S. [EuroQol-5D: a simple alternative for measuring health-related quality of life in primary care]. Aten Primaria. 2001 Oct 15;28(6):425-30. doi: 10.1016/s0212-6567(01)70406-4. No abstract available. Spanish. PMID 11602124
- [Background] Guillen-Riquelme A, Buela-Casal G. [Psychometric revision and differential item functioning in the State Trait Anxiety Inventory (STAI)]. Psicothema. 2011 Aug;23(3):510-5. Spanish. PMID 21774907
- [Background] Spielberger CD, Gorsuch RL, Lushene RE. Cuestionario de ansiedad estado-rasgo. Madrid: Tea. 1982;1.
- [Background] Lopez MA, Gabilondo A, Codony M, Garcia-Forero C, Vilagut G, Castellvi P, Ferrer M, Alonso J. Adaptation into Spanish of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) and preliminary validation in a student sample. Qual Life Res. 2013 Jun;22(5):1099-104. doi: 10.1007/s11136-012-0238-z. Epub 2012 Jul 27. PMID 22836376
- [Background] Castellvi P, Forero CG, Codony M, Vilagut G, Brugulat P, Medina A, Gabilondo A, Mompart A, Colom J, Tresserras R, Ferrer M, Stewart-Brown S, Alonso J. The Spanish version of the Warwick-Edinburgh mental well-being scale (WEMWBS) is valid for use in the general population. Qual Life Res. 2014 Apr;23(3):857-68. doi: 10.1007/s11136-013-0513-7. Epub 2013 Sep 5. PMID 24005886
- [Background] Royuela Rico A, Macías Fernández JA. Propiedades clinimetricas de la versión castellana del cuestionario de Pittsburgh. Vigilia-Sueño [Internet]. 1997;9(2):81-94. Available from: https://www.researchgate.net/publication/258705863
- [Background] Miller K, Feucht W, Schmid M. Bioactive Compounds of Strawberry and Blueberry and Their Potential Health Effects Based on Human Intervention Studies: A Brief Overview. Nutrients. 2019 Jul 2;11(7):1510. doi: 10.3390/nu11071510. PMID 31269727